CLINICAL TRIAL: NCT01825434
Title: Effect of Yogurt Containing Polydextrose, Lactobacillus Acidophilus NCFM and Bifidobacterium Lactis HN019: a Randomized, Double-blind, Controlled Study in Chronic Constipation
Brief Title: Effect of Yogurt With Polydextrose,L Acidophilus and B Lactis in Chronic Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Claudio Saddy Rodrigues Coy, PhD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE 454/2008
Record Dates: First submitted 2013-02-26; First posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-01

CONDITIONS: Constipation
Keywords: chronic constipation; Lactobacillus acidophilus NCFM; Bifidobacterium lactis HN019
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Active Comparator): yogurt containing polydextrose, L. acidophilus NCFM® (ATCC 700396) and B. lactis HN019 (AGAL NM97/09513) 1 time per day, for 30 days.
  Interventions: Dietary Supplement: yogurt containing: polydextrose L. acidophilus NCFM® B. lactis HN019
- Placebol group (Placebo Comparator): regular yogurt, 1 time per day for 30 days.

INTERVENTIONS:
Dietary Supplement: yogurt containing: polydextrose L. acidophilus NCFM® B. lactis HN019 — NCFM Group
  Other Names: acidophilus NCFM® (ATCC 700396); lactis HN019 (AGAL NM97/09513)
  Arms: Treatment Group

SUMMARY:
Background and aims:Constipation is a frequent complaint and the combination of a prebiotic and probiotics would have a potentially synergic effect on the intestinal transit. The present study therefore aims to investigate the combination of polydextrose (Litesse®), L. acidophilus NCFM® and B. lactis HN019 in a yogurt on intestinal transit in subjects who suffer from constipation.

Methods: Patients with constipation were randomly divided into two groups, Placebo Group (PG) and Treatment Group (TG), and had to eat 180 ml of unflavored yogurt every morning for 14 days. Those in the CG received only yogurt, while the TG received yogurt containing polydextrose, L. acidophilus NCFM® (ATCC 700396) and B. lactis HN019 (AGAL NM97/09513). Expect that patients who took a combination of polydextrose has a decrease in the colonic transit time (CTT) when comparing initial and final transit time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chonic constipation
* agachan between 10 and 20
* bowel transit time with ingestion of 24 radiopaque markers (Sitzmarks) and retention of 80% of them on day 5

Exclusion Criteria:

* Patients with hypothyroidism
* antidepressant users
* normal colonic
* transit time (24 hrs or less) as well as higher than 96 hours were

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Colonic transit | Colonic transit time and Agachan score will be evaluated before and in day15 aftler yogurt ingestion. All particIpants will be followed for 30 days after the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Claudio SR Coy, Ph.D, Study Chair — University of Campinas, Brazil
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil